CLINICAL TRIAL: NCT04356586
Title: Immune Response to Covid-19 in 300 Health Care Workers With Mild Symptoms
Status: Completed | Type: Observational
Sponsor: Sciensano (Other Government)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Maria Gpossens, Scientific collaborator, Sciensano
Other Study IDs: Jessa300
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: COVID-19; Serology
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Three hundred healthcare workers with mild symptoms for Covid-19 will be followed during three months. Each two weeks, serological tests will be performed. Re-infection will be monitored by saliva-swabs.

ELIGIBILITY:
Inclusion Criteria:

* HCW previous tested for Covid-19 with mild symptoms in Jessa Ziekenhuis, Belgium

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HCW previous tested for Covid-19 with mild symptoms in Jessa Ziekenhuis, Belgium
Sampling Method: Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Percentage of serological positive healthcare workers | three months
Percentage of HCW with positive Saliva-sabs | three months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Goossens, MD, PhD, Principal Investigator — Sciensano
Locations (1):
- Sciensano, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No